CLINICAL TRIAL: NCT07175324
Title: Correlation Between Optical Coherence Tomography Angiography and Visual Field Changes in Patients With Multiple Sclerosis
Brief Title: Oct-A and Perimetry in Multiple Sclerosis
Acronym: MS
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Gamal Nouby Mahmoud, Doctor, Assiut University
Other Study IDs: OctA in Multiple sclerosis
Record Dates: First submitted 2025-09-03; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: MS; OctA
MeSH Terms: conditions — Multiple Sclerosis | interventions — Visual Field Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with multiple sclerosis
  Interventions: Device: optical coherence tomography angiography; Device: Visual Field Perimetry
- healthy control
  Interventions: Device: optical coherence tomography angiography; Device: Visual Field Perimetry

INTERVENTIONS:
Device: optical coherence tomography angiography — correlation between OctA and Visual field changes in Multiple Sclerosis
Device: Visual Field Perimetry — Correlation between OctA and Visual field changes in Multiple sclerosis

SUMMARY:
This study aims to assess retinal vascular density using OCT-A and correlate these parameters with visual field changes in MS patients with and without a history of ON

DETAILED DESCRIPTION:
The aim of this work is to investigate the correlation between visual field parameters and optical coherence tomography angiography (OCT-A) findings in patients with multiple sclerosis (MS). MS is a chronic autoimmune demyelinating disease that frequently involves the visual pathway, often presenting with optic neuritis (ON) and subsequent neurodegeneration. OCT-A, a non-invasive imaging modality, enables detailed visualization and quantification of retinal microvasculature, particularly the superficial and deep capillary plexuses, which supply the retinal ganglion cells and nerve fiber layers. Previous studies have demonstrated reduced retinal vessel density and thinning of retinal nerve fiber layer (RNFL) and ganglion cell complex (GCC) in MS patients, reflecting neuro-axonal damage and microvascular impairment. However, the relationship between these structural and vascular changes and functional visual outcomes, such as visual field loss, remains to be fully elucidated.

This study aims to assess retinal vascular density using OCT-A and correlate these parameters with visual field indices in MS patients with and without a history of ON. By analyzing inter-eye differences and comparing with MS patients, the research seeks to clarify whether OCT-A metrics can serve as reliable biomarkers for visual dysfunction and disease progression in MS. Understanding this correlation could improve early detection of neuroretinal damage, guide monitoring of disease activity, and potentially inform therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting multiple sclerosis (RR-MS) or other MS subtypes confirmed by established neurological criteria. .Ability to undergo OCTA imaging and visual field testing. .Visual acuity sufficient to perform reliable visual field testing.
* Absence of other ocular diseases affecting the retina or optic nerve (e.g., diabetic retinopathy, glaucoma)

Exclusion Criteria:

.History of ocular diseases unrelated to MS that could confound OCTA or visual field results.

.Recent optic neuritis episode within a defined period (often 3-6 months) to avoid acute inflammation effects.

.Media opacities preventing quality OCTA imaging. .Systemic diseases that may affect retinal vasculature (e.g., uncontrolled hypertension, diabetes).

.Poor cooperation or inability to complete visual field testing reliably

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with multiple sclerosis and healthy control group in Assiut
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
1-To evaluate the correlation between OCTA-derived microvascular metrics {Structural measure} and visual field defects{Functional measure} in patients with multiple sclerosis (MS) | baseline
  The aim of this work is to investigate the correlation between visual field parameters and optical coherence tomography angiography (OCT-A) findings in patients with multiple sclerosis (MS). MS is a chronic autoimmune demyelinating disease that frequently involves the visual pathway, often presenting with optic neuritis (ON) and subsequent neurodegeneration. OCT-A, a non-invasive imaging modality, enables detailed visualization and quantification of retinal microvasculature, particularly the superficial and deep capillary plexuses, which supply the retinal ganglion cells and nerve fiber layers. Previous studies have demonstrated reduced retinal vessel density and thinning of retinal nerve fiber layer (RNFL) and ganglion cell complex (GCC) in MS patients, reflecting neuro-axonal damage and microvascular impairment. However, the correlation between these structural and vascular changes and functional visual outcomes, such as visual field loss, remains to be fully elucidated.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mancino, R., Martucci, A., Di Costanzo, A., et al. (2021).Optical coherence tomography and optical coherence tomography angiography findings in multiple sclerosis patientshttps://www.tandfonline.com/doi/full/10.1080/01658107.2021.1963787
- [Background] Liu J, Song S, Gu X, Li H, Yu X. Microvascular impairments detected by optical coherence tomography angiography in multiple sclerosis patients: A systematic review and meta-analysis. Front Neurosci. 2023 Jan 13;16:1121899. doi: 10.3389/fnins.2022.1121899. eCollection 2022. PMID 36711144
- [Background] Farci R, Carta A, Cocco E, Frau J, Fossarello M, Diaz G. Optical coherence tomography angiography in multiple sclerosis: A cross-sectional study. PLoS One. 2020 Jul 23;15(7):e0236090. doi: 10.1371/journal.pone.0236090. eCollection 2020. PMID 32702050
- [Background] Mohammadi S, Gouravani M, Salehi MA, Arevalo JF, Galetta SL, Harandi H, Frohman EM, Frohman TC, Saidha S, Sattarnezhad N, Paul F. Optical coherence tomography angiography measurements in multiple sclerosis: a systematic review and meta-analysis. J Neuroinflammation. 2023 Mar 27;20(1):85. doi: 10.1186/s12974-023-02763-4. PMID 36973708